CLINICAL TRIAL: NCT04347291
Title: Mobile Phone Support for Adults and Support Persons to Live Well With Diabetes
Acronym: FAMS 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Lindsay Mayberry, Principal Investigator, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 200398; R01DK119282 (NIH)
Record Dates: First submitted 2020-03-30; First posted 2020-04-15 (Actual); Results first posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes
Keywords: family support; social support; text message; mobile health; hemoglobin A1c
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The investigators use mail-in A1c kits for the primary outcome - hemoglobin A1c - and the lab analyzing these samples is masked to study description or participants' assigned condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FAMS 2.0 (Experimental): Patient participants will receive FAMS 2.0 components (monthly phone coaching and text message support for goals and medication adherence) for nine months. Linked support persons will receive text message support tailored to the goal set by the patient participant.
  All patient participants will receive text messages advising how to access their study A1c test results, and receive high-quality print materials including a book upon enrollment and quarterly newsletters on healthy living with diabetes. All support person participants will receive high-quality print materials including a book and information about providing quality social support upon enrollment and quarterly newsletters on healthy living with diabetes.
  Interventions: Behavioral: FAMS 2.0; Behavioral: Print Materials
- Print Materials (Placebo Comparator): All patient participants will receive text messages advising how to access their study A1c test results, and receive high-quality print materials including a book upon enrollment and quarterly newsletters on healthy living with diabetes. All support person participants will receive high-quality print materials including a book and information about providing quality social support upon enrollment and quarterly newsletters on healthy living with diabetes.
  Interventions: Behavioral: Print Materials

INTERVENTIONS:
Behavioral: FAMS 2.0 — FAMS components include monthly phone coaching following a semi-structured protocol plus daily automated text message support to the patient participant and less frequent automated text messages to their support person, if enrolled.
  Other Names: Family/friend Activation to Motivate Self-care; (prior iteration) Family-focused Add-on to Motivate Self-care (NCT02481596)
  Arms: FAMS 2.0
Behavioral: Print Materials — Quality print materials about diabetes management provided upon enrollment and in quarterly study newsletters.

SUMMARY:
This study evaluates a mobile phone-delivered intervention (FAMS 2.0; Family/friend Activation to Motivate Self-care) designed to help adults with type 2 diabetes set and achieve self-care goals and improve the quality of family/friend support for their goals. The investigators hypothesize that FAMS 2.0 will improve glycemic control and reduce diabetes distress among patients and reduce support burden and diabetes distress in enrolled support persons. The investigators hypothesize the mechanisms by which FAMS 2.0 will affect these outcomes for the patient include (a) increased helpful and reduced harmful family/friend involvement, (b) increased self-care (i.e., diet, physical activity, medication adherence), and (c) increased diabetes self-efficacy.

DETAILED DESCRIPTION:
The 9-month FAMS 2.0 intervention is an expansion and improvement of a previously evaluated intervention (FAMS; NCT02481596). FAMS components include:

* Monthly coaching sessions (20-30 minutes each) with patient participants by phone focusing on helpful/unhelpful/desired family and friend behaviors relevant to the patients' self-identified diet, exercise, and/or stress management goal
* Daily one-way and interactive text messages to the patient to support him/her in meeting the identified daily goal and medication adherence
* Weekly interactive text messages asking the patient to reflect on goal progress followed by personalized feedback from the coach
* The option to invite an adult support person to receive text messages (3 one-way per week and one interactive text per week) encouraging the support person to discuss the patient's self-care goal to provide opportunities for the patient to practice skills discussed during phone coaching

Participants will be randomized in a parallel design to either FAMS 2.0 or an active control. Our target enrollment is N=334 dyads (patient participants and support persons). Patients are encouraged to invite a support person, but it is not required. Patients and their support person will be randomized together (if enrolled). The study is powered to detect a 0.5% reduction in hemoglobin A1c. Analyses will examine effects at 9 months (post-intervention) and 15 months (sustained effects). The investigators will impute missing data, including all participants completing at least two data collection periods in analyses. Participants will be analyzed as randomized regardless of withdrawal from the intervention (i.e., intention-to-treat principals).

ELIGIBILITY:
Inclusion Criteria:

PATIENTS:

* Speaks and reads in English
* 18-75 years old
* Diagnosed with type 2 diabetes
* Receiving outpatient care from a partnering clinic
* Community dwelling (e.g., not in a nursing facility)
* Prescribed at least one daily diabetes medication
* Owns a mobile phone

SUPPORT PERSONS:

* Speaks and reads in English
* 18 years or older
* Owns a mobile phone

Exclusion Criteria:

PATIENTS:

* Unable to communicate by phone
* Pregnant currently
* Currently undergoing treatment for cancer (e.g., radiation, chemotherapy)
* Diagnosed with end-stage renal disease
* Receiving hospice services
* Diagnosed with congestive heart failure
* Diagnosed with dementia
* Diagnosed with schizophrenia
* Reported current abuse during screening
* Demonstrates inability to receive and respond to a text
* Does not take medication on his/her own/medication administered by someone else

SUPPORT PERSONS:

- Demonstrates inability to receive and respond to a text

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 638 (Actual)
Dates: Start 2020-04-28 (Actual); Primary Completion 2023-02-17 (Actual); Study Completion 2023-02-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
After study results are posted on clinical trials and published, de-identified data will be available upon requests made to the principal investigator.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After study results are posted on clinical trials and outcomes published in a peer-reviewed journal, until 5 years later.
Access Criteria: Contact the principal investigator

REFERENCES:
- [Derived] Roddy MK, Spieker AJ, Greevy RA Jr, Nelson LA, Berg C, Mayberry LS. Diabetes-specific family functioning typology associated with intervention engagement and effects: secondary analyses from a randomized controlled trial. Ann Behav Med. 2025 Jan 4;59(1):kaae070. doi: 10.1093/abm/kaae070. PMID 39661957
- [Derived] Roddy MK, El-Rifai M, LeStourgeon L, Aikens JE, Wolever RQ, Greevy RA, Mayberry LS. Prerandomization withdrawals from a Type 2 diabetes self-care support intervention trial are associated with lack of available support person coparticipant. Chronic Illn. 2025 Mar;21(1):105-114. doi: 10.1177/17423953231203734. Epub 2023 Sep 26. PMID 37750180
- [Derived] Mayberry LS, El-Rifai M, Nelson LA, Parks M, Greevy RA Jr, LeStourgeon L, Molli S, Bergner E, Spieker A, Aikens JE, Wolever RQ. Rationale, design, and recruitment outcomes for the Family/Friend Activation to Motivate Self-care (FAMS) 2.0 randomized controlled trial among adults with type 2 diabetes and their support persons. Contemp Clin Trials. 2022 Nov;122:106956. doi: 10.1016/j.cct.2022.106956. Epub 2022 Oct 5. PMID 36208719

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We recruited patient participants with a goal of 334 enrolled. Patient participants could invite a support person to enroll with them, but this was not required. 638 represents 338 patient participants and 300 support persons.
Pre-assignment Details: 9 patient participants were administratively withdrawn prior to randomization; 6 of those participants also had a support person enrolled who was administratively withdrawn. These patient participants were unreachable during a pre-determined run-in period after enrollment and therefore withdrawn per protocol.
Groups:
- FAMS 2.0: Patient participants will receive FAMS 2.0 components (monthly phone coaching and text message support for goals and medication adherence) for nine months. Linked support persons will receive text message support tailored to the goal set by the patient participant.
  All patient participants will receive text messages advising how to access their study A1c test results, and receive high-quality print materials including a book upon enrollment and quarterly newsletters on healthy living with diabetes. All support person participants will receive high-quality print materials including a book and information about providing quality social support upon enrollment and quarterly newsletters on healthy living with diabetes.
  FAMS 2.0: FAMS components include monthly phone coaching following a semi-structured protocol plus daily automated text message support to the patient participant and less frequent automated text messages to their support person, if enrolled.
  Print Materials: Quality print materials about diabetes management provided upon enrollment and in quarterly study newsletters.
Period: Overall Study
Arm/Group | FAMS 2.0 | Print Materials
Started (Patient participants were randomized with their support person (if enrolled), but support person participation was not required. There were 294 patient/support person dyads (329 patient participants, 294 support persons; 35 patients participated without a support person).) | 314 | 309
Patient Participants | 164 | 165
Support Persons | 150 | 144
Completed | 304 | 297
Not Completed | 10 | 12

BASELINE CHARACTERISTICS:
Population: Patient participants had the option to invite a support person, but support person participation was not required. Patient participants were randomized with their support person (if enrolled). There were 329 patient participants and 294 support persons (294 patient/support person dyads; 35 patients participated without a support person).
Groups:
- Total: Total of all reporting groups
Arm/Group | FAMS 2.0 | Print Materials | Total
Number analyzed (Participants) | 314 | 309 | 623
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Patient participants were randomized with their support person (if enrolled). There were 329 patient participants and 294 support persons (294 patient/support person dyads; 35 patients participated without a support person).
  years
    Patient participants: number analyzed (Participants) | 164 | 165 | 329
    Patient participants | 56.1 (11.0) | 57.9 (10.5) | 57.0 (10.8)
    Support persons: number analyzed (Participants) | 150 | 144 | 294
    Support persons | 50.4 (14.7) | 53.4 (14.0) | 51.9 (14.4)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Patient participants were randomized with their support person (if enrolled). There were 329 patient participants and 294 support persons (294 patient/support person dyads; 35 patients participated without a support person)..
  Participants
    Patient participants: number analyzed (Participants) | 164 | 165 | 329
    Patient participants: Male | 85 | 85 | 170
    Patient participants: Female | 77 | 80 | 157
    Patient participants: Prefer to self-describe | 2 | 0 | 2
    Patient participants: Unknown or not reported | 0 | 0 | 0
    Support persons: number analyzed (Participants) | 150 | 144 | 294
    Support persons: Male | 42 | 38 | 80
    Support persons: Female | 102 | 103 | 205
    Support persons: Prefer to self-describe | 0 | 0 | 0
    Support persons: Unknown or not reported | 6 | 3 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Patient participants were randomized with their support person (if enrolled). There were 329 patient participants and 294 support persons (294 patient/support person dyads; 35 patients participated without a support person).
  Participants
    Patient participants: number analyzed (Participants) | 164 | 165 | 329
    Patient participants: Hispanic or Latino | 13 | 12 | 25
    Patient participants: Not Hispanic or Latino | 151 | 152 | 303
    Patient participants: Unknown or Not Reported | 0 | 1 | 1
    Support persons: number analyzed (Participants) | 150 | 144 | 294
    Support persons: Hispanic or Latino | 8 | 6 | 14
    Support persons: Not Hispanic or Latino | 135 | 132 | 267
    Support persons: Unknown or Not Reported | 7 | 6 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Patient participants were randomized with their support person (if enrolled). There were 329 patient participants and 294 support persons (294 patient/support person dyads; 35 patients participated without a support person).
  Participants
    Patient participants: number analyzed (Participants) | 164 | 165 | 329
    Patient participants: American Indian or Alaska Native | 0 | 0 | 0
    Patient participants: Asian | 8 | 8 | 16
    Patient participants: Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
    Patient participants: Black or African American | 35 | 44 | 79
    Patient participants: White | 115 | 105 | 220
    Patient participants: More than one race | 3 | 3 | 6
    Patient participants: Unknown or Not Reported | 2 | 4 | 6
    Support persons: number analyzed (Participants) | 150 | 144 | 294
    Support persons: American Indian or Alaska Native | 1 | 0 | 1
    Support persons: Asian | 8 | 6 | 14
    Support persons: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Support persons: Black or African American | 30 | 36 | 66
    Support persons: White | 97 | 92 | 189
    Support persons: More than one race | 5 | 2 | 7
    Support persons: Unknown or Not Reported | 9 | 8 | 17
Hemoglobin A1c (patient participants) [Mean (Standard Deviation); unit: percent] — Hemoglobin A1c assessed by mail-in A1c kits from CoreMedica and/or taken from electronic health record (venipuncture or point-of-care) Population: Hemoglobin A1c data was collected from patient participants (n=329) and used in the analysis of the primary outcome measure.
  percent
    number analyzed (Participants) | 164 | 165 | 329
    (all) | 8.64 (1.79) | 8.53 (1.56) | 8.59 (1.68)
Diabetes distress (patient participants) [Mean (Standard Deviation); unit: score on a scale] — as assessed by the Problem Areas in Diabetes (PAID-5) with scores ranging 0-100 where higher scores indicate more distress (worse) Population: Patient participants' diabetes distress was assessed at baseline and used in the analysis of the primary outcome measure. There were 329 patient participants.
  score on a scale
    number analyzed (Participants) | 164 | 165 | 329
    (all) | 38.8 (26.9) | 38.1 (24.5) | 38.5 (25.7)
Psychosocial well-being (patient participants) [Mean (Standard Deviation); unit: score on a scale] — as assessed by the World Health Organization - Five Well-Being Index (WHO-5) with scores ranging 0 to 100 where higher scores indicate more well-being (better) Population: Patient participants' psychosocial well-being was assessed at baseline and used in the analysis of the primary outcome measure. There were 329 patient participants.
  score on a scale
    number analyzed (Participants) | 164 | 165 | 329
    (all) | 55.6 (23.4) | 56.5 (23.1) | 56.1 (23.2)

OUTCOME MEASURES:

1. Primary Outcome: Change in Glycemic Control (Patient Participants) During Intervention Period
Description: Hemoglobin A1c assessed by mail-in A1c kits from CoreMedica and/or taken from electronic health record (venipuncture or point-of-care) where higher values indicate worse glycemic control
Time Frame: Baseline and 6 and 9 months post-baseline
Population: Patient participants
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 164 | 165
percent
  Baseline | 8.64 (1.79) | 8.53 (1.56)
  6 months | 8.00 (1.55) | 8.31 (1.55)
  9 months | 8.23 (1.72) | 8.05 (1.41)

2. Primary Outcome: Change in Glycemic Control (Patient Participants) Sustained Post-intervention Effects
Description: as for outcome 1
Time Frame: Baseline and 12 and 15 months post-baseline
Population: Patient participants
Measure: Mean (Standard Deviation); unit: percent
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 164 | 165
percent
  Baseline | 8.64 (1.79) | 8.53 (1.56)
  12 months | 7.99 (1.55) | 8.04 (1.41)
  15 months | 8.21 (1.62) | 8.04 (1.40)

3. Primary Outcome: Change in Diabetes Distress (Patient Participants) During Intervention Period
Description: Assessed by the Problem Areas in Diabetes (PAID-5) with scores ranging 0-100 where higher scores indicate more distress (worse)
Time Frame: Baseline and 6 and 9 months post-baseline
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 164 | 165
score on a scale
  Baseline | 38.8 (26.9) | 38.1 (24.5)
  6 months | 30.1 (25.4) | 32.9 (24.8)
  9 months | 26.5 (25.4) | 30.6 (22.8)

4. Primary Outcome: Change in Diabetes Distress (Patient Participants) Sustained Post-intervention Effect
Description: as for outcome 3
Time Frame: Baseline and 15 months post-baseline
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 164 | 165
score on a scale
  Baseline | 38.8 (26.9) | 38.1 (24.5)
  15 months | 26.2 (25.5) | 27.8 (22.4)

5. Primary Outcome: Change in Psychosocial Well-being (Patient Participants) During Intervention Period
Description: Assessed by the World Health Organization - Five Well-Being Index (WHO-5) with scores ranging 0 to 100 where higher scores indicate more well-being (better)
Time Frame: Baseline and 6 and 9 months post-baseline
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 164 | 165
score on a scale
  Baseline | 55.6 (23.4) | 56.5 (23.1)
  6 months | 62.5 (23.2) | 57.5 (22.9)
  9 months | 62.2 (22.2) | 61.4 (22.2)

6. Primary Outcome: Change in Psychosocial Well-being (Patient Participants) Sustained Post-intervention Effect
Description: as for outcome 5
Time Frame: Baseline and15 months post-baseline
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 164 | 165
score on a scale
  Baseline | 55.6 (23.4) | 56.5 (23.1)
  15 months | 62.0 (23.1) | 65.3 (23.0)

7. Secondary Outcome: Change in Diabetes Distress (Support Person Participants) During Intervention Period
Description: as assessed by the Problem Areas in Diabetes (PAID-5) Family Member Version. Scores range 0-100 where higher scores indicate more diabetes distress experienced by the support person (worse)
Time Frame: Baseline and 6 and 9 months post-baseline
Population: Support person participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 150 | 144
score on a scale
  Baseline | 34.2 (22.2) | 31.4 (21.6)
  6 months | 31.9 (22.4) | 28.4 (20.1)
  9 months | 30.2 (21.8) | 28.3 (22.2)

8. Secondary Outcome: Change in Diabetes Distress (Support Person Participants) Sustained Post-intervention Effect
Description: Assessed by the Problem Areas in Diabetes (PAID-5) Family Member Version. Scores range 0-100 with higher scores indicate more diabetes distress experienced by the support person (worse)
Time Frame: Baseline and 15 months post-baseline
Population: Support person participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 150 | 144
score on a scale
  Baseline | 34.2 (22.2) | 31.4 (21.6)
  15 months | 28.9 (22.5) | 27.8 (20.7)

9. Secondary Outcome: Change in Support Burden (Support Person Participants) During Intervention Period
Description: as assessed by the Impact of Diabetes Profile-Family Members from the Diabetes Attitudes Wishes and Needs Study-2 (DAWN2). Scores range 0 to 4 where higher scores indicate greater support burden (worse)
Time Frame: Baseline and 6 and 9 months post-baseline
Population: Support person participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 150 | 144
score on a scale
  Baseline | 0.392 (0.760) | 0.360 (0.674)
  6 months | 0.341 (0.690) | 0.368 (0.746)
  9 months | 0.392 (0.710) | 0.366 (0.716)

10. Secondary Outcome: Change in Support Burden (Support Person Participants) Sustained Post-intervention Effect
Description: as assessed by the Impact of Diabetes Profile-Family Members from the Diabetes Attitudes Wishes and Needs Study-2 (DAWN2). Scores range 0 to 100 where higher scores indicate greater support burden (worse)
Time Frame: Baseline and 15 months post-baseline
Population: Support person participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 150 | 144
score on a scale
  Baseline | 0.392 (0.760) | 0.360 (0.674)
  15 months | 0.301 (0.664) | 0.368 (0.750)

11. Other Pre Specified Outcome: Change in Diabetes Self-efficacy (Patient Participants - Outcome & Mediator)
Description: as assessed by the Perceived Diabetes Self-Management Scale with scores ranging 8 to 40 with higher scores indicating more self-efficacy (better)
Time Frame: Baseline and 6 and 9 months post-baseline
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 164 | 165
score on a scale
  Baseline | 25.7 (6.74) | 25.0 (6.41)
  6 months | 29.6 (6.85) | 26.4 (6.74)
  9 months | 30.2 (6.65) | 27.8 (6.50)

12. Other Pre Specified Outcome: Change in Dietary Behavior (Patient Participants - Outcome & Mediator)
Description: as assessed by Personal Diabetes Questionnaire, Use of Information for Decision Making Scale with scores ranging 1-6 where higher scores indicate more use of dietary information for decision making (better)
Time Frame: Baseline and 6, 9, and 15 months post-baseline
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 164 | 165
score on a scale
  Baseline | 3.00 (1.53) | 3.15 (1.48)
  6 months | 3.43 (1.61) | 3.40 (1.45)
  9 months | 3.64 (1.49) | 3.37 (1.43)
  15 months | 3.30 (1.43) | 3.31 (1.42)

13. Other Pre Specified Outcome: Change in Dietary Behavior (Patient Participants - Outcome & Mediator)
Description: as assessed by Personal Diabetes Questionnaire, Problem Eating Behavior scale with scores ranging 1-6 where higher scores indicate more problem eating behaviors (worse)
Time Frame: Baseline and 6, 9, and 15 months post-baseline
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 164 | 165
score on a scale
  Baseline | 3.73 (1.09) | 3.78 (0.983)
  6 months | 3.23 (0.898) | 3.58 (1.01)
  9 months | 3.19 (0.919) | 3.43 (1.07)
  15 months | 3.29 (1.02) | 3.44 (1.08)

14. Other Pre Specified Outcome: Change in Physical Activity (Patient Participants - Outcome & Mediator)
Description: as assessed by a modified Rapid Assessment of Physical Activity with scores ranging 0 to 6533 with higher scores indicating more physical activity (better)
Time Frame: Baseline and 6, 9, and 15 months post-baseline
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 164 | 165
score on a scale
  Baseline | 670 (840) | 830 (969)
  6 months | 873 (943) | 782 (982)
  9 months | 890 (1146) | 789 (1020)
  15 months | 782 (957) | 777 (941)

15. Other Pre Specified Outcome: Change in Diabetes Medication Adherence (Patient Participants - Outcome & Mediator)
Description: as assessed by the Summary of Diabetes Self-Care Activities medications subscale with scores ranging 0 to 7 representing days in the prior week with perfect adherence (higher better)
Time Frame: Baseline and 6, 9, and 15 months post-baseline
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 164 | 165
score on a scale
  Baseline | 6.22 (1.55) | 6.22 (1.48)
  6 months | 6.56 (1.12) | 6.38 (1.46)
  9 months | 6.39 (1.57) | 6.29 (1.54)
  15 months | 6.44 (1.33) | 6.48 (1.14)

16. Other Pre Specified Outcome: Change in Diabetes Medication Adherence (Patient Participants - Outcome & Mediator)
Description: as assessed by the Adherence to Refills and Medications in Diabetes scale, with scores ranging 11-44 with higher scores indicating more problems with adherence (worse)
Time Frame: Baseline and 6, 9, and 15 months post-baseline
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 164 | 165
score on a scale
  Baseline | 15.3 (4.38) | 14.9 (3.36)
  6 months | 13.9 (3.41) | 14.3 (3.27)
  9 months | 13.7 (3.20) | 14.3 (3.66)
  15 months | 14.1 (3.75) | 14.2 (3.87)

17. Other Pre Specified Outcome: Change in Helpful Diabetes-specific Family/Friend Involvement (Patient Participants - Outcome & Mediator)
Description: as assessed by the Helpful Involvement scale of Family/friend Involvement in Adults' Diabetes with scores ranging 1 to 5 with higher scores indicating more helpful involvement (better)
Time Frame: Baseline and 6, 9, and 15 months post-baseline
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 164 | 165
score on a scale
  Baseline | 2.33 (1.04) | 2.27 (1.04)
  6 months | 2.86 (1.06) | 2.28 (1.07)
  9 months | 2.74 (1.14) | 2.33 (1.01)
  15 months | 2.48 (1.05) | 2.34 (1.06)

18. Other Pre Specified Outcome: Change in Helpful Diabetes-specific Family/Friend Involvement (Patient Participants - Outcome & Mediator)
Description: as assessed by the Important Others Climate Questionnaire, specific to diabetes management, with scores ranging 1 to 5 with higher scores indicating more autonomy supportive communication (better)
Time Frame: Baseline and 6, 9, and 15 months post-baseline
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 164 | 165
score on a scale
  Baseline | 3.45 (0.870) | 3.50 (0.871)
  6 months | 3.81 (0.804) | 3.58 (0.961)
  9 months | 3.79 (0.865) | 3.58 (0.947)
  15 months | 3.66 (0.954) | 3.49 (0.962)

19. Other Pre Specified Outcome: Change in Harmful Diabetes-specific Family/Friend Involvement (Patient Participants - Outcome & Mediator)
Description: as assessed by the Harmful Involvement scale of Family/friend Involvement in Adults' Diabetes with scores ranging 1 to 5 with higher scores indicating more harmful involvement (worse)
Time Frame: Baseline and 6, 9, and 15 months post-baseline
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 164 | 165
score on a scale
  Baseline | 1.66 (0.547) | 1.67 (0.630)
  6 months | 1.62 (0.588) | 1.62 (0.621)
  9 months | 1.53 (0.589) | 1.55 (0.532)
  15 months | 1.54 (0.516) | 1.60 (0.649)

20. Other Pre Specified Outcome: Change in Harmful Diabetes-specific Family/Friend Involvement (Patient Participants - Outcome & Mediator)
Description: as assessed by the criticism items from the Family Emotional Involvement and Criticism Scale, specific to diabetes management, with scores ranging 0 to 16 with higher scores indicating more perceived criticism (worse)
Time Frame: Baseline and 6, 9, and 15 months post-baseline
Population: Patient participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 164 | 165
score on a scale
  Baseline | 4.15 (4.06) | 3.52 (3.42)
  6 months | 3.26 (3.59) | 3.11 (3.40)
  9 months | 3.00 (3.57) | 2.82 (3.30)
  15 months | 2.87 (3.28) | 3.10 (3.56)

21. Other Pre Specified Outcome: Change in Helpful Support Person Involvement (Support Person Participants - Outcome & Mediator)
Description: as assessed by the Helpful Involvement scale of Family/friend Involvement in Adults' Diabetes - support person version. Scores ranging 1 to 5 with higher scores indicating more helpful involvement (better)
Time Frame: Baseline and 6, 9, and 15 months post-baseline
Population: Support person participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 150 | 144
score on a scale
  Baseline | 2.66 (0.946) | 2.53 (1.03)
  6 months | 3.11 (1.01) | 2.47 (0.947)
  9 months | 3.04 (0.988) | 2.49 (0.997)
  15 months | 2.74 (0.974) | 2.37 (0.921)

22. Other Pre Specified Outcome: Change in Harmful Support Person Involvement (Support Person Participants - Outcome & Mediator)
Description: as assessed by the Harmful Involvement scale of Family/friend Involvement in Adults' Diabetes - support person version. Scores ranging 1 to 5 with higher scores indicating more harmful involvement (worse)
Time Frame: Baseline and 6, 9, and 15 months post-baseline
Population: Support person participants
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 150 | 144
score on a scale
  Baseline | 1.50 (0.439) | 1.49 (0.492)
  6 months | 1.38 (0.448) | 1.38 (0.453)
  9 months | 1.39 (0.472) | 1.39 (0.472)
  15 months | 1.37 (0.368) | 1.35 (0.443)

23. Other Pre Specified Outcome: Change in Support Person Involvement Alignment (Support Person Participants - Outcome & Mediator)
Description: as assessed by items from the Family Experience of Patient Involvement measure from the Diabetes Attitudes Wishes and Needs Study-2 (DAWN2). Scores range 0 to 4 where a score of 2 indicates alignment between the support person's current level of involvement and their desired level of involvement. We will report change in the % aligned (reporting a 2) across conditions.
Time Frame: Baseline and 6, 9, and 15 months post-baseline
Population: Support person participants
Measure: Count of Participants; unit: Participants
Arm/Group | FAMS 2.0 | Print Materials
Number analyzed (Participants) | 150 | 144
Participants
  Baseline | 46 | 44
  6 months | 67 | 70
  9 months | 65 | 65
  15 months | 65 | 69

ADVERSE EVENTS:
Time Frame: We followed participants for 15 months of study participation, with the first participant enrollment in April 2020 until the last participant completed 15-month follow-up in February 2023.
Groups:
- FAMS 2.0-Patient Participants; FAMS 2.0-Support Persons: Patient participants will receive FAMS 2.0 components (monthly phone coaching and text message support for goals and medication adherence) for nine months. Linked support persons will receive text message support tailored to the goal set by the patient participant.
  All patient participants will receive text messages advising how to access their study A1c test results, and receive high-quality print materials including a book upon enrollment and quarterly newsletters on healthy living with diabetes. All support person participants will receive high-quality print materials including a book and information about providing quality social support upon enrollment and quarterly newsletters on healthy living with diabetes.
  FAMS 2.0: FAMS components include monthly phone coaching following a semi-structured protocol plus daily automated text message support to the patient participant and less frequent automated text messages to their support person, if enrolled.
  Print Materials: Quality print materials about diabetes management provided upon enrollment and in quarterly study newsletters.
- Print Materials-Patient Participants; Print Materials-Support Persons: All patient participants will receive text messages advising how to access their study A1c test results, and receive high-quality print materials including a book upon enrollment and quarterly newsletters on healthy living with diabetes. All support person participants will receive high-quality print materials including a book and information about providing quality social support upon enrollment and quarterly newsletters on healthy living with diabetes.
  Print Materials: Quality print materials about diabetes management provided upon enrollment and in quarterly study newsletters.
Arm/Group | FAMS 2.0-Patient Participants | FAMS 2.0-Support Persons | Print Materials-Patient Participants | Print Materials-Support Persons
All-Cause Mortality (participants affected / at risk) | 1/164 | 0/150 | 2/165 | 0/144
Serious Adverse Events (participants affected / at risk) | 0/164 | 0/150 | 0/165 | 0/144
Other Adverse Events (participants affected / at risk) | 0/164 | 0/150 | 0/165 | 0/144

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-10-24): https://cdn.clinicaltrials.gov/large-docs/91/NCT04347291/Prot_001.pdf
  • Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/91/NCT04347291/SAP_002.pdf
  • Informed Consent Form (2021-03-25): https://cdn.clinicaltrials.gov/large-docs/91/NCT04347291/ICF_000.pdf